CLINICAL TRIAL: NCT03659656
Title: Fight Hypertension in the Digital Age
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Yang Bai, Assistant Professor, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-0051
Record Dates: First submitted 2018-08-28; First posted 2018-09-06 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Pre Hypertension; Hypertension
MeSH Terms: conditions — Prehypertension; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fitbit (FB) (Other): The Fitbit only (FB) group will receive the Fitbit monitor to use for 3 months.
  Interventions: Device: Fitbit usage
- Fitbit + Health coaching (FB+) (Experimental): The Fitbit + Health coaching (FB+) group will receive a Fitbit, weekly personalized physical activity report and health coaching by phone. The 3-month intervention will be delivered through health coaching (1-time per week for month 1, 1-time every other week for month 2 and 1 time for month 3) and use of a Fitbit activity monitor.
  Interventions: Behavioral: Lifestyle coaching; Device: Fitbit usage

INTERVENTIONS:
Behavioral: Lifestyle coaching — Goal setting and behavior change barriers will be discussed through lifestyle behavioral change coaching. Personalized weekly physical activity achievement report will also be sending to participants in experimental group. The participants will also have a Fitbit to use for 3 months.
  Other Names: Fitbit Charge HR
  Arms: Fitbit + Health coaching (FB+)
Device: Fitbit usage — The participants will have a Fitbit to use for 3 months.

SUMMARY:
The estimated prevalence of hypertension is approximately 29.0% in the United States during 2015-2016. Hypertension remains an important public health challenge in the United States because it increases the risk for other health conditions such as cardiovascular disease. Strong evidence has indicated that physical activity is associated with reduced risk of hypertension. Lifestyle change programs, including physical activity promotion and dietary modification, have been shown to effectively reduce the cumulative incidence of hypertension for individuals at-risk. However, it is challenging to maintain a high-level program. Recently, the consumer marketplace has been flooded with an array of wearable activity monitors, such Fitbit and Apple Watch, designed to enhance real time self-assessment and activity behavior change. These devices provide potential to serve as more cost effective and appealing intervention means for behavior change applications. Studies have examined the accuracy of the devices but little has been done to examine the monitors' feasibility as a behavior change strategy in and of themselves or as an adjunct to traditional methods (e.g., education and goal setting through a health coach), among people with hypertension. The real-time physical activity monitoring also provides an opportunity to build customized physical activity biofeedback for behavior change. Thus, there is an increasing interest to investigate their application as a behavior change strategy in isolation or as a complement to a more traditional intervention. The current study will recruit participants with hypertension and pre-hypertension. A Fitbit Charge HR will be provided to use over the intervention to all participants. They will be randomly assigned into Fitbit only and Fitbit plus (adding weekly personalized report and health coach consulting) groups for 3-months.

DETAILED DESCRIPTION:
After potential participants contact the research team, the research team will schedule a phone screening with them to make sure they meet the criteria. If they pass the phone screening, visit 1 will be scheduled. If they fail the phone screening, their contact information and response to the phone screening questions will be destroyed. If an individual agrees to participate, they will complete the informed consent and they will be assigned a unique ID number. Eligibility will be first checked. Blood pressure will be measured three times using an automated blood pressure cuff after participants have been seated and rested for at least 10 minutes for an accurate reading. For participants who do not take medication that managing blood pressure, if they have systolic blood pressure <120mmHg or diastolic blood pressure <80mmHg they will not be allowed to participate. If an individual has systolic blood pressure >140mmHg or diastolic blood pressure >90mmHg they will not be allowed to participate without approval from their physician. If they are diagnosed with pre-hypertension or hypertension and are currently taking medication, they will need to provide a physician's note to participate. They will also be asked to complete a physical activity measure, the International Physical Activity Questionnaire (IPAQ) to assess their activity over the last week. If they accumulated more than 150 minutes of moderate and vigorous physical activity per week, they will not be eligible to participate. This will be checked by a member of the research team to ensure that they are eligible to participate. If the person meets criteria (other inclusion and exclusion criteria information is listed below separately in Inclusion/Exclusion section), they will be provided with additional information about the study and be guided through the Visit 1 data collection protocol and be informed about plans for Visit 2 (1 week later) and Visit 3 (approximately 3 months later). The visits will last about 60 minutes each, with Visit 2 being up to 90 minutes for participants randomly assigned to the Fitbit + Behavior Change Strategies (FB+) condition described below.

Visit 1. Visit 1 will include baseline measurements and providing participants with information about the monitors that they will wear to assess physical activity and sedentary behaviors at baseline and at the end of the intervention. They will schedule a time to come back the following week for their second study visit.

Visit 2. At the beginning of Visit 2, participants will be block randomized to their experimental condition and informed of their condition assignment. Randomization will occur in blocks of 5 to ensure that groups are experiencing similar environmental (e.g. weather) variations that may influence physical activity behaviors. Randomization will be done using a random number generator. Conditions are: use of the Fitbit alone (FB) or use of the Fitbit in combination with behavior change strategies (FB+). Descriptions of conditions are below. Regardless of condition, all participants will receive information about the Fitbit and will be given a guided tour of the device itself and the associated software. Participants will be given a username and password to be used with the software and will be encouraged to utilize the software over the next 3 months to assist them in becoming more physically active. Participants assigned to the FB condition will use their Fitbit on their own for the duration of 3-month intervention, similar to the experience of participants buying the device off-the-shelf. Those assigned to the FB+ condition will discuss their perceived benefits and barriers of becoming more physically active with health coach. Participants will also be encouraged to set a goal of their choosing related to using their Fitbit to increase their physical activity. Weekly progress reports will be sent to participants through Email on Monday. Participants assigned to this group will also receive weekly (first month), semi-monthly (second month), monthly (third month) phone contact from the health coach to follow-up on the achievement from previous week(s) and re-evaluate their goals based on their current behaviors.

Regardless of group assignment, during the 3-month intervention all participants will receive periodic (~monthly) contacts (via email or phone) from the research team asking how they are using their Fitbits. For participants in the FB+ group, this contact can be at the same time as their check-ins. During this monthly contact, participants will be asked open-ended questions regarding how frequently the Fitbits are being worn, how often participants are looking at their data, and what aspects of the monitors and associated software/apps are particularly useful and/or motivating for them. They will be also asked about their physical health and well beings related to participate in the study as a safety check.

Approximately one week prior to the final visit (~3 months after the start of the intervention), participants will be asked to come to the lab for a brief visit to pick up an objective activity monitor (ActiGraph) and to wear them for the next week in order to assess physical activity and sedentary time at the end of the intervention. At this time, participants will also be scheduled to return for their final study visit.

Visit 3 will be completed at the end of the 3-month trial. During this visit, participants will complete the same anthropomorphic, cardiovascular, and psychosocial measures assessed at baseline. They will be given the opportunity to complete an optional semi-structured interview with a member of the study team. This brief interview could be done during this visit or at another time that is convenient for the participant. The purpose of the interview would be to gather qualitative information from participants regarding their use of the monitors and factors that facilitated and/or impeded behavior change.

Twelve weeks after the intervention the investigator's will ask participants to complete the physical activity questionnaire once again to assess for long term changes in self-reported physical activity and secondary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 24-60.
* Willing to wear a Fitbit monitor for a period of 3 months.
* Able to read and speak English.
* Have a computer and/or smartphone and internet access to be able to make use of the Fitbit.
* Pre- and/or hypertension: systolic blood pressure >120mmHg or diastolic blood pressure >80mmHg. Not taking medication: If an individual has systolic blood pressure >140mmHg or diastolic blood pressure >90mmHg they will not be allowed to participate without approval from their physician. Currently taking medication: they will need to provide a physician's note to participate.
* Inactive: less than 150 min/week of exercise over the past 3 months and not currently participating in a structured exercise program.

Exclusion Criteria:

* Individuals who are currently using a Fitbit or similar monitoring device to track their physical activity.
* Individuals with injuries or conditions that prevent them from safely participating in physical activity
* cardiovascular or cerebrovascular disease
* Cancer, requiring treatment in the past 5 years
* Other medical condition that is life-threatening or can interfere with or be aggravated by participating in physical activity

Ages: 24 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline daily steps and moderate and vigorous physical activity minutes at 3 months | The primary outcome will be measured twice, one at baseline and another one at approximately one week prior to the final visit (~3 months after the start of the intervention).
  Daily steps and moderate and vigorous physical activity minutes will be measured by ActiGraph GT3X+ for 7 days at the baseline and post-intervention at 3 months.

SECONDARY OUTCOMES:
Change from baseline self-efficacy (sticking to it and making time for exercise) | The secondary outcome will be measured twice, one at baseline and another one at the end of 3 months intervention.
  Self-efficacy for exercise will be assessed at the baseline and post-intervention at 3 months.There are two scales of this survey, Sticking to it and Making time for exercise. The range of two scales are 1 to 5. Higher values represent better outcome.
Change from baseline self-regulation (time-management, goal-setting, relapse prevention, self-monitoring, reinforcement, and social support) | The secondary outcome will be measured twice, one at baseline and another one at the end of 3 months intervention.
  Six aspects of self-regulation are measured with the Physical Activity Self-Regulation instrument (PASR-12) including time-management, goal-setting, relapse prevention, self-monitoring, reinforcement, and social support. The instrument contains 12 measures on a 5 point Likert-type scale ranging from 1=never to 5=very often. The self-regulation score is calculated as the sum of the 12 responses. The minimum possible score is 12 and the maximum possible score is 60 with a higher score indicating more frequent use of self-regulation strategies for participation in physical activity.
Change from baseline social support (family participation, family rewards and punishment, and friend participation) | The secondary outcome will be measured twice, one at baseline and another one at the end of 3 months intervention.
  Social support for exercise will be measured using the "Social Support and Exercise Survey," a 13-item questionnaire to measure three factors: family participation, family rewards and punishment, and friend participation. Answers range from 1-5 representing none, rarely, a few times, often, and very often or "does not apply." The potential score ranges from 10-50 for both family participation and friend participation, and from 3-15 for family rewards and punishment for a total potential score of 23-115.
Change from baseline self-motivation | The secondary outcome will be measured twice, one at baseline and another one at the end of 3 months intervention.
  Self-motivation for exercise will be measure using 'Self-Motivation Inventory', a 40-item questionnaires with answers range from 1-5. The potential score ranges from 40-200, with a high score indicative of high self-motivation.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Bai, PhD, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: Undecided